CLINICAL TRIAL: NCT05163470
Title: Effectiveness of a New On Field Rehabilitation Framework for Return to Sport in Injured Elite Football Players - a Prospective Randomized Controlled Trial
Brief Title: On Field Functional Rehabilitation -Comparing Two Programs-framework
Acronym: FIREframework
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dr. Konstantinos Fousekis, Ass.Professor in Sports Physical Therapy, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: statioan1906198402833125882688
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Sport Injury
Keywords: football; Return to sports; injuries; On filed functional rehabilitation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The population of the study will be divided randomized in two groups, each of the group it will follow a different functional on field rehabilitation framework in low limb musculoskeletal injuries after sustain an acute injury.The two groups will be divided in subgroups,each of group with the same division ,based on the nature of musculoskeletal injury.A physician,will evaluate the players on initial time of the acute injury and after the compliancy of the rehabilitation.Each of the functional on field rehabilitation framework will be applied from one physiotherapist.All the subject will receive the same physiotherapy treatment ,i.e. manual therapy and specific therapeutic exercise protocol depending of the nature of the injury.After return to sports all the participants will be follow the same prevention program depending of the nature of the injury for two months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On Fi.RE. framework (Experimental): Men football professional players
  Interventions: Other: early on filed functional rehabilitation
- Traditional rehabilitation (Active Comparator): Men football professional players
  Interventions: Other: traditional on filed functional rehabilitation

INTERVENTIONS:
Other: early on filed functional rehabilitation — Intervention 1 ,called ''On FI.RE. framework '' included a on filed functional rehabilitation framework ,with early return of the player on the field activities during injury recovery. Involve a specific 5 stages framework of functional rehabilitation on filed. Criteria of inclusion and exclusion for each stage are included based on pain, oedema and range of motion specific to nature of injury . Additional included a daily session planning framework for on field functional rehabilitation with a content ,duration and the description of each content.
  Arms: On Fi.RE. framework
Other: traditional on filed functional rehabilitation — Intervention 2 ,called 'traditional rehabilitation' include a on field functional rehabilitation framework ,as the late phase of injury recovery .The framework described as a 5 stages on filed rehabilitation framework based on load monitoring usingGlobal positioning system.No criteria for the player to return to activity on the field cited ,but referred criteria for progression in each stage based on Strength/power depending of the nature of injury.
  Arms: Traditional rehabilitation

SUMMARY:
Background Nowadays, in elite demanding football, injuries are a delicate issue as affects player's availability for the teams to win games and attain trophies.Following an injury, the appropriate recovery is vital to return athletes quickly and safely to their sport, based on pre injury physical and psychological levels. Delay in rehabilitation can result in prolonged pain and a delayed return to sports, a finding that emphasizes the importance of proper rehabilitation procedure during injury recovery.On field functional rehabilitation, a key point in injury recovery in football , as presented in the definition of rehabilitation ,obtained the interaction of the person with the environment he lives and provide him/her the ability to optimize functionality. Especially in sports, the last one is applied via ecological theory in sports with a wealth of benefits for the player during injury recovery on filed. Ecological theory bring us closer to the sport from a realistic approach , can provide an explanation to many situations that arise in sports and understands the athlete as a part of his/her own surroundings.

Ideally, through injury recovery , the focus should be more on the biological time needed for the injury to recover, while trying to maintain the skills of the athlete during the rehabilitation process. Adequate and appropriate cognitive and neuromuscular skills should be maintained in high level, in activities that normally occurred during training or games. In this Context, application of ecological theory in football on field functional rehabilitation provide to the player the ability to maintain this skills, according with the high demands of elite football players.The maximum retention of football specific skills and the adaptation of injured tissue in an injury football player take place on his/her natural environment of action , the field .

What sports medicine community knows? Until today, disunity of opinions prevalent among sports medicine community about on filed functional rehabilitation during injury recovery.The majority of the clinicians apply on field functional rehabilitation, called as traditional on filed rehabilitation, as the late phase of injury recovery ,where the player comeback on filed activity when he had already restore maximum or the average strength and function based on pre injury screening or standard value.The progression of the player during the late phase of injury recovery based on load monitoring with (global position system) to control progression and risk of reinjury. On the contrary emphasized the opinion of the early return to filed activity that's can increase for the injury player the ability to maintain sports specific skills as much as he can during injury recovery.

In the literature review there is a absence of evidence to refer to a specific framework for on field functional rehabilitation in regard of recovery an injured football player (elite or amateur ) on field. References ,with a lack of evidence ,exist only in some specific rehabilitation protocols such as muscle injury rehabilitation tendons injuries management or Anterior Cruciate Ligament Reconstruction rehabilitation as the late phase of injury recovery.Only one study, present on field functional rehabilitation framework of 5 stages based on traditional rehabilitation for short and long term injuries based on load monitoring through global position system ,as a work based on experience and lacking of evidence.

Aim The overall objective of the proposed research is to conduct a prospective randomized controlled trial to evaluate the effectiveness of ''On FI.RE. framework'' (on filed rehabilitation framework),namely the early return to on field activities during an injury recovery. Included a specific 5 stages program-framework , and a daily session planning framework for on field functional rehabilitation. The effectiveness will evaluated with the time that the player needed to return to full participation in teams training.

DETAILED DESCRIPTION:
Background Nowadays, in elite demanding football, injuries are a delicate issue as affects player's availability for the teams to win games and attain trophies. Injury was defined, using a time-loss definition, as any physical complaint sustained by a player that results from a football match or football training and led to the player being unable to take full part in future football training or match.An elite football team, constituted from about 25 players, presented an injury incident of 6.6./1000 hours of exposure, (decreased 3% the last years) . Following an injury, the appropriate recovery is vital to return athletes quickly and safely to their sport, based on pre injury physical and psychological levels. Delay in rehabilitation can result in prolonged pain and a delayed return to sports, a finding that emphasizes the importance of proper rehabilitation procedure during injury recovery .

Rehabilitation is defined as a set of interventions designed to optimize function and reduce disability in individuals with healthy conditions in interaction with their environment.This interaction refers to the observation of animals , so in fact the person, as the animals, has the ability to execute an action or movement based on the environment he lives.The last one is applied in ecological theory in sports with a wealth of benefits for the player during training or injury recovery on filed. Ecological theory bring us closer to the sport from a realistic approach , can provide an explanation to many situations that arise in sports,understands the athlete as a part of his/her own surroundings where there is only perception and action and also presented the large degree of freedom that can exist in a movement which surpasses the conscious capacity of control in nervous system.

Ideally, through injury recovery , the focus should be more on the biological time needed for the injury to recover, while trying to maintain the skills of the athlete during the rehabilitation process.Adequate and appropriate cognitive and neuromuscular skills should be maintained in high level, in activities that normally occurred during training or games. In this Context, application of ecological theory in football on field functional rehabilitation provide to the player the ability to maintain this skills, according with the high demands of elite football players.The successful persistence of athlete skills during injury rehabilitation and decision making process will come through neuroplasticity which exerts an important role and allows to correct, modify, and adapt neuromuscular patterns, allowing the athlete to protect the injured part during the biological time needed for it to heal and to maintain the sports skills.This would allow adaption and healing of the injured tissue, restoring as quickly as possible the specific movements or loads expected from the injured muscle or joint.The maximum retention of football specific skills and the adaptation of injured tissue in an injury football player take place on his/her natural environment of action , the field.

What sports medicine community knows? Until today, disunity of opinions prevalent among sports medicine community about on filed functional rehabilitation during injury recovery.The majority of the clinicians apply on field functional rehabilitation, called as traditional on filed rehabilitation, as the late phase of injury recovery ,where the player comeback on filed activity when he had already restore maximum or the average strength and function based on pre injury screening or standard value.The progression of the player during the late phase of injury recovery based on load monitoring with global position system to control progression and risk of reinjury.In oone study traditional rehabilitation is described and analyzed more specifically as the overlap period between the rehabilitation and return to sports .On the contrary emphasized that the early return to filed activity for the injury player to maintain sports specific skills as much as he can during injury recovery.

In the literature review there is a absence of evidence to refer to a specific framework for on field functional rehabilitation in regard of recovery an injured football player (elite or amateur ) on field. References ,with a lack of evidence ,exist only in some specific rehabilitation protocols such as muscle injury rehabilitation tendons injuries management or Anterior Cruciate Ligament Reconstruction rehabilitation as the late phase of injury recovery. In one study, presented on field functional rehabilitation framework of 5 stages based on traditional rehabilitation for short and long term injuries based on load monitoring through global position system as a work based on experience and lacking of evidence.

Aim The overall objective of the proposed research is to conduct a prospective randomized controlled trial to evaluate the effectiveness of ''On FI.RE. framework'' (on filed rehabilitation framework),namely the early return to on field activities during an injury recoveryIncluded a specific 5 stages program-framework , and a daily session planning framework for on field functional rehabilitation. The effectiveness will be evaluated with the time that the player will be needed to return to full participation in teams training.

Protocol The eligible study population will consist of men professional football players that participate in Greek football professional categories ,between 17-40 years old ,with an acute low limb musculoskeletal injury that sustained in game or training. Participants of the study will be divided in two groups. One group will be treated with 'On FI.RE. framework' during on field functional rehabilitation and the other group(control group)will be treated with 'traditional rehabilitation' framework. Each group will be categorized in subgroups based on the nature of injury such as muscle tear, ligament tear, acute overuses syndromes and fractures or cartilage lesions. All players fulfilling the inclusion and not meeting the exclusion criteria will be asked to participate in the study. After the player´s enrolment has been confirmed and informed consent is obtained a set of questionnaires is provided for background data on medical history based on football federation medical examination paper. A physician will make the evaluation and diagnostic imaging prescription to make a diagnosis of the injury . When the procedure is completed, the patient is randomized. One physiotherapist, different for each group, will apply the general(physiotherapy and exercises in the Gym) and specific(on filed functional rehabilitation) program. The intervention program analyzed in chapter 8. If a player don't complete or quit from the procedure he will withdraw for the data collection. After the completion of the rehabilitation program the physician will evaluate the player to permit or not, the full participation in team training. After the return of player's to team training will follow a secondary prevention program for two months. Participation in this study will last maximum twelve months.

Statistical analysis plan To address the primary and secondary objectives, a statistical analysis by using statistical package for the social sciences will be performed. Depending on the data distribution ,a X² test or Mann-Whitney U test will be applied to calculate the means between the two groups based on time player needed to return in team training.

The importance of the presented study lie on the presentation and development of evidence in clinical practice regarding the ideal of on field functional rehabilitation framework ,for low limb musculoskeletal injuries for professional football players in the matter of faster and safety return to play.

ELIGIBILITY:
Inclusion Criteria:

* Subject/player he will be a professional player at least 3 years
* The musculoskeletal injury to be an acute injury
* The player participate in the study from the initial tine that injury occurred
* The injury to be moderate or severe (≥ 7 days ) as the initial diagnosis (1)

Exclusion Criteria:

* A reinjury of a previous injury
* Chronic overuse syndrome or other disorders that affect the intervention and the result of the study
* Do not sustained another injury the last two months

Ages: 17 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure is time to return, that is, time that the player needed from injury to full participation in the team training process based on pre injury physical level. | Direct after rehabilitation completion
  Time to return ,namely loss days ,is defined as the period of absence for a player following an injury constituted the full period (number of days) between the date when the player was forced to discontinue his football participation due to an injury until the date when the medical team allowed the player to return to full participation in team training.After the completion of the measurement , means of the total number of days that players of each group needed to return to full participation in team training will be compared between groups to evaluate which of the two interventions is more effective.
Time to return-subgroups | Direct after rehabilitation completion
  After the completion of the measurement , means of the total number of days that players of each subgroup (based on th nature of injury) needed to return to full participation in team training will be compared between subgroups of two arms to evaluate which of the two interventions is more effective.

SECONDARY OUTCOMES:
Occurrence of reinjuries, injury of the same type and at the same site as an index injury, was registered during a 2 month period after the player return to performance. | For nine months after Return to sports
  ''Early recurrence'' ,a recurrent injury occurring within 2 months of a player's return to full participation and ''late recurrence'' a recurrent injury occurring 2 to 12 months after a player's return to full participation,with the team in games will be documented. The result it will be compared between groups .

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Stathas, Bachelor, Study Chair — student of MSc therapeutic exercise
Locations (3):
- Greece (3):
  - Stadium of Agios Nikolaos, Agios Nikolaos, Crete
  - Hymettus Municipal Stadium, Athens, Imittos
  - Municipal Stadium of Aigion, Aigio, Peloponnese

IPD SHARING:
Plan to Share IPD: No
The subjects are professional football players and their data aren't permitted to be published

REFERENCES:
- [Background] Ekstrand J, Krutsch W, Spreco A, van Zoest W, Roberts C, Meyer T, Bengtsson H. Time before return to play for the most common injuries in professional football: a 16-year follow-up of the UEFA Elite Club Injury Study. Br J Sports Med. 2020 Apr;54(7):421-426. doi: 10.1136/bjsports-2019-100666. Epub 2019 Jun 10. PMID 31182429
- [Background] Ekstrand J, Spreco A, Bengtsson H, Bahr R. Injury rates decreased in men's professional football: an 18-year prospective cohort study of almost 12 000 injuries sustained during 1.8 million hours of play. Br J Sports Med. 2021 Oct;55(19):1084-1091. doi: 10.1136/bjsports-2020-103159. Epub 2021 Feb 5. PMID 33547038
- [Background] Buckthorpe M, Frizziero A, Roi GS. Update on functional recovery process for the injured athlete: return to sport continuum redefined. Br J Sports Med. 2019 Mar;53(5):265-267. doi: 10.1136/bjsports-2018-099341. Epub 2018 Sep 29. No abstract available. PMID 30269097
- [Background] Bizzini M, Hancock D, Impellizzeri F. Suggestions from the field for return to sports participation following anterior cruciate ligament reconstruction: soccer. J Orthop Sports Phys Ther. 2012 Apr;42(4):304-12. doi: 10.2519/jospt.2012.4005. Epub 2012 Mar 30. PMID 22467065
- [Background] Buckthorpe M, Della Villa F, Della Villa S, Roi GS. On-field Rehabilitation Part 2: A 5-Stage Program for the Soccer Player Focused on Linear Movements, Multidirectional Movements, Soccer-Specific Skills, Soccer-Specific Movements, and Modified Practice. J Orthop Sports Phys Ther. 2019 Aug;49(8):570-575. doi: 10.2519/jospt.2019.8952. Epub 2019 Jul 10. PMID 31291556
- [Background] Della Villa S, Boldrini L, Ricci M, Danelon F, Snyder-Mackler L, Nanni G, Roi GS. Clinical Outcomes and Return-to-Sports Participation of 50 Soccer Players After Anterior Cruciate Ligament Reconstruction Through a Sport-Specific Rehabilitation Protocol. Sports Health. 2012 Jan;4(1):17-24. doi: 10.1177/1941738111417564. PMID 23016064
- [Background] Taberner M, Allen T, Cohen DD. Progressing rehabilitation after injury: consider the 'control-chaos continuum'. Br J Sports Med. 2019 Sep;53(18):1132-1136. doi: 10.1136/bjsports-2018-100157. Epub 2019 Feb 8. No abstract available. PMID 30737202
- [Background] Fuller CW, Ekstrand J, Junge A, Andersen TE, Bahr R, Dvorak J, Hagglund M, McCrory P, Meeuwisse WH. Consensus statement on injury definitions and data collection procedures in studies of football (soccer) injuries. Br J Sports Med. 2006 Mar;40(3):193-201. doi: 10.1136/bjsm.2005.025270. PMID 16505073
- [Derived] Stathas I, Kalliakmanis A, Kekelekis A, Danassi Afentaki D, Tsepis E, Fousekis K. Effectiveness of an On-Field Rehabilitation framework for return to sports in injured male professional football players: a single-blinded, prospective, randomised controlled trial. BMJ Open Sport Exerc Med. 2024 Jan 19;10(1):e001849. doi: 10.1136/bmjsem-2023-001849. eCollection 2024. PMID 38268525
- See also: Information, affordances, and the control of action in sport — http://www.ijsp-online.com/abstract/view/40/79